CLINICAL TRIAL: NCT03930784
Title: A Real-world Study to Examine the Relationship Between Simple Physical Functioning Tests, Complications and Recovery Following Abdominal Surgery - a Prospective Cohort Study
Brief Title: A Real-world Study to Examine the Relationship Between Simple Physical Functioning Tests, Complications and Recovery Following Abdominal Surgery.
Status: Completed | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Collaborators: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, mary flahive, Senior Physiotherapist, Practice Tutor, University Hospital of Limerick
Other Study IDs: 043/16
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Surgery--Complications; Abdomen; Physical Activity
Keywords: physical function; recovery; abdominal
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Divided for analysis as having suffered post-operative complications or not
  Interventions: Other: Nil intervention

INTERVENTIONS:
Other: Nil intervention

SUMMARY:
Background: Complications impact physical and psychological recovery and are associated with financial cost. General physical function has not been studied in relation to the development of surgical complications in this cohort.

Objective: Evaluate the physical function performance differences between those who develop complications and those who do not and determine their impact on recovery.

Design: Observational Setting: The pre-operative assessment unit in the University Hospital Limerick. Patients: Forty-nine participants who were planned to undergo abdominal surgery were recruited & 43 completed the study.

Main outcome measure: Demographics, physical function, lung function, surgical parameters, complications and recovery data was collected.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Eighteen years or above
* Planned for elective abdominal surgery
* American Society of Anaesthesia physical status score <4.

Exclusion Criteria:

* Abdominal surgery within one year prior to study entry
* Unable or unwilling to give informed consent
* Inability (cognitive) to perform the pre-operative tests, as characterised by inability to understand the information in the patient information leaflet
* Current systemic acute illness
* Scheduled for non-abdominal surgery
* Unstable angina or myocardial infarction in the previous month
* Physical limitation precluding inability to participate in pre-operative tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants scheduled to under-go elective abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with complications & changes over time points. | (1) 0-29 days, (2) 30 and (3) 60 days post operatively
  Defined as occuring within the first 30 days post-operatively using the Clavien Dindo classification

SECONDARY OUTCOMES:
Spirometry to measure lung function | 2-4 weeks pre-operatively
  Spirometry was performed to obtain the participant's vital capacity, forced vital capacity, forced expiratory pressure in one second ratio and peak expiratory flow rate.
  The instructions and methods used were as per the American Thoracic Society Guidelines 2005. Testing required participants to perform two different tests, three times each. In the initial test, participants were seated and instructed to inhale as deeply as possible before blowing into the spirometer until they felt they needed to inhale again. The second test required them to be seated and after a maximal inhalation, to exhale as forcefully as they could until they felt the need to inhale again. Results were recorded numerically and as a percentage compared to norms of the same sex, race, age, and height. This data was generated by the spirometer (Vitalograph Model 2120 Hand Held REF 79XXX) post testing.
Peak Cough Flow to measure cough strength | 2-4 weeks pre-operatively
  This was performed by attaching a naso-oral mask to a peak flow meter (Mini- Wright Peak Flow Meter, Clement Clarke International). Figure 2.5. Participants were requested to inhale maximally, in a seated position, prior to placing the mask over their nose and mouth, and coughing forcefully. This was repeated three times to give numerical scores. The highest score was recorded. New face masks and flow meters were used for each patient. Results were recorded in litres per minute (L/min). The researcher attempted to limit any reliability bias by using standardised instructions and corrections as required.
Six Minute Walk Test to measure exercise capacity | 2-4 weeks pre-operatively
  This was performed as per the ATS guidelines 2002, as recommended by Biccard 2005. Participants were instructed to walk up and down a thirty-metre distance, over a six-minute period, and each length was recorded. The thirty-metre distance was measured with each metre marked, and the same area used for each test. If they were not at a start or endpoint at the six-minute mark, the distance that they had covered was recorded. Predicted distance was calculated against normative data based on age, sex, weight and height. Participants peak oxygen uptake (VO2Peak) was also calculated as per Ross et al 2010.
Thirty Second Sit to Stand Test to measure endurance | 2-4 weeks pre-operatively
  Participants were asked to go from a seated to standing position and vice versa, as many times as possible in thirty seconds, without the use of their hands to assist. The same standard height chair (17 inches) was used throughout which was placed against a wall for safety. Participants were instructed by the researcher when to start and stop, using a standard stopwatch. When the clock reached thirty seconds, if they were more than half way to a full stand, this was regarded as a stand.Results were recorded as numerical data.
Grip strength. | 2-4 weeks pre-operatively
  Grip strength was recorded, using a Baseline hydraulic hand held dynamometer, as a measure of overall physical function, independent of lower limb strength.Participants were asked to squeeze the dynamometer maximally for a period of 3 seconds, the result was recorded and the test repeated twice more. An average of the scores was recorded in pounds (lbs).
Change over time in activity levels. | (1) 2-4 weeks pre-operatively, (2) 30 and (3) 60 days post operatively
  This data was collected by the researcher using the short form International Physical Activity Questionnaire (IPAQ) which is a self-reported measure of activity levels in the previous seven days (IPAQ Research Committee 2005). The IPAQ incorporates questions relating to vigorous and moderate activities, as-well as walking and sitting time. It uses patient subjective reports to quantify the time spent, if any, doing the previously mentioned activities in the previous week. The patients weekly metabolic equivalents (METS) were then calculated using the formula and descriptors provided in the scoring protocol.Sedentary time was calculated in weekly minutes by multiplying their daily minutes answers by seven.
Changes in perceived recovery over time | 30 and 60 days post operatively
  Participants were asked to self-assess their own physical recovery using the same questions and classification as used in a study by Onerupp et al 2015.

IPD SHARING:
Plan to Share IPD: No